CLINICAL TRIAL: NCT01164410
Title: The Efficacy Side Effects and the Tolerance of Polyethylene Glycol 3350 as a Bowel Prep in Children
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CCF 09-378
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Colonoscopy: Patients undergoing colonoscopy in the Department of Pediatric Gastroenterology at the Cleveland Clinic Children's Hospital in Cleveland, Ohio.

SUMMARY:
Bowel preparation solutions containing Polyethylene Glycol is a commonly used preparation of the colon for colonoscopy in children. However young children and adolescents often subject to the volume and taste of liquid that must be consumed for an adequate preparation. Currently almost all of our patients experience some difficulty with completing the colyte preparation and approximately 10-20% is unable to achieve adequate cleansing due to inability to drink the solution. The standard colyte solution is salty and often impedes children from drinking the required amount of colyte preparation for adequate colon cleansing. Miralax has been used at a dose of 1.5gm/kg/day to a maximum of 102 gms /day as four day prep Four day bowel prep can be extremely frustrating for the parents and the patients. This may result in low patient acceptance, limiting compliance leading to inadequate colonoscopy. Decreasing the duration of the prep may increase the compliance and provide better colon visualization.

Hence a Cross sectional study looking at the safety,efficacy,tolerability of PEG 3350 mixed in Gatorade G(TM) as a bowel prep in children needs to be conducted. Consent will be obtained from parents and assent will be obtained from patients. Previous laboratory tests for each patient will be reviewed. All patients in the study will be required to consume MiralaxTM/Gatorade GTM the day prior to their procedure. The patients will be given written instructions as to how to much solution to take and how to prepare and consume the solution. The patient shall be maintained on a clear liquid diet the day prior to the procedure. Once patients arrive for the colonoscopy they will be asked to complete a questionnaire regarding their bowel preparation. Prior to the administration of IV fluids, 1ml of blood will be obtained a basic metabolic panel. The patient will then undergo a colonoscopy by routine procedure and technique. The endoscopist will complete a questionnaire when done with the colonoscopy to rate the cleanliness of the colon.

We propose that MiralaxTM combined with Gatorade GTM given the day prior to colonoscopy is a safe, tolerable and efficacious cleansing regimen for colonoscopy in children.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Patients five years old or older that present to the pediatric GI clinic and are capable of taking oral liquids and have been scheduled for a colonoscopy.
2. Patients who are able to communicate their discomfort and preferences.

Exclusion Criteria:

1. Patients that are neurologically compromised
2. Patients in need of emergent colonoscopy
3. Patients with known metabolic, endocrine, renal or cardiac conditions.
4. Presence of pre-existing ostomy, short bowel syndrome, gastric retention, intestinal obstruction or swallowing difficulties.
5. Patients with known electrolyte abnormalities.
6. Patients who are allergic to PEG-3350.
7. Patients that are known to be pregnant.
8. Patients with known fructose intolerance.
9. Patient younger than five years old.

ELIGIBILITY:
Inclusion Criteria:

* Patients five years old or older that present to the pediatric GI clinic and are capable of taking oral liquids and have been scheduled for a colonoscopy.
* Patients who are able to communicate their discomfort and preferences.

Exclusion Criteria:

* Patients that are neurologically compromised
* Patients in need of emergent colonoscopy
* Patients with known metabolic, endocrine, renal or cardiac conditions.
* Presence of pre-existing ostomy, short bowel syndrome, gastric retention, intestinal obstruction or swallowing difficulties.
* Patients with known electrolyte abnormalities.
* Patients who are allergic to PEG-3350.
* Patients that are known to be pregnant.
* Patients with known fructose intolerance.
* Patient younger than five years old.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Forty-five patients undergoing colonoscopy in the Department of Pediatric Gastroenterology at the Cleveland Clinic Children's Hospital in Cleveland, Ohio.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
MiralaxTM combined with Gatorade GTM given the day prior to colonoscopy is a safe, tolerable and efficacious cleansing regimen for colonoscopy in children. | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Childrens Hospital, Cleveland, Ohio, United States